CLINICAL TRIAL: NCT01847274
Title: A Phase 3 Randomized Double-blind Trial of Maintenance With Niraparib Versus Placebo in Patients With Platinum Sensitive Ovarian Cancer.
Brief Title: A Maintenance Study With Niraparib Versus Placebo in Patients With Platinum Sensitive Ovarian Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tesaro, Inc. (Industry)
Collaborators: European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other); Myriad Genetics, Inc. (Industry); US Oncology Research (Industry); Sarah Cannon (Industry); Cooperative Ovarian Cancer Group (COGI) (Unknown); Facing Our Risk of Cancer Empowered (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 213356; PR-30-5011-C (Other: Tesaro)
Record Dates: First submitted 2013-04-11; First posted 2013-05-06 (Estimated); Results first posted 2019-05-01 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Ovarian Neoplasms; Platinum Sensitive Ovarian Cancer
Keywords: ovarian cancer; platinum sensitive; gBRCAmut; BRCA; high-grade serous histology; PARP inhibitor
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Niraparib (Active Comparator): 2:1 Ratio administered once daily continuously during a 28 day cycle.
  Interventions: Drug: Active comparator: Niraparib
- Placebo (Placebo Comparator): Administered once daily continuously over a 28 day cycle.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Active comparator: Niraparib — Niraparib vs placebo 2:1 ratio
  Other Names: Niraparib
  Arms: Niraparib
Drug: placebo
  Arms: Placebo

SUMMARY:
This is a Phase 3, multicenter, randomized, double-blind, placebo-controlled study of niraparib as maintenance in platinum sensitive ovarian cancer patients who have either gBRCAmut or a tumor with high-grade serous histology and who have responded to their most recent chemotherapy containing a platinum agent. Niraparib is an orally active PARP inhibitor. Niraparib or placebo (in a 2:1 ratio) will be administered once daily continuously during a 28-day cycle. Health-related quality of life will be measured by the Functional Assessment of Cancer Therapy - Ovarian Symptom Index (FOSI), European Quality of Life scale, 5-Dimensions (EQ-5D), and a neuropathy questionnaire. Safety and tolerability will be assessed by clinical review of adverse events (AEs), physical examinations, electrocardiograms (ECGs), and safety laboratory values.

The primary objective of this study is to evaluate efficacy of niraparib as maintenance therapy in patients who have platinum sensitive ovarian cancer as assessed by the prolongation of progression free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, female, any race
* Histologically diagnosed ovarian cancer, fallopian tube cancer or primary peritoneal cancer
* High grade (or grade 3) serous histology or known to have gBRCAmut
* Has received at least 2 previous courses of platinum-containing therapy, and has disease that was considered platinum sensitive following the penultimate (next to last) platinum course (more than 6 month period between penultimate platinum regimen and progression of disease)
* Has responded to last the platinum regimen, remains in response and is enrolled on study within 8 weeks of completion of the last platinum regimen
* ECOG 0-1
* Adequate bone marrow, kidney and liver function

Exclusion Criteria:

* Known hypersensitivity to the components of niraparib
* Invasive cancer other than ovarian cancer within 2 years (except basal or squamous cell carcinoma of the skin that has been definitely treated)
* Symptomatic uncontrolled brain metastasis
* Is pregnant or breast feeding
* Immunocompromised patients
* Known active hepatic disease
* Prior treatment with a known PARP inhibitor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Actual)
Dates: Start 2013-06-21 (Actual); Primary Completion 2016-04-22 (Actual); Study Completion 2021-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Studies, Study Director — GlaxoSmithKline
Locations (97):
- United States (30):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Palo Alto, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Burlington, Massachusetts
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Morristown, New Jersey
  - GSK Investigational Site, Farmington, New Mexico
  - GSK Investigational Site, Lake Success, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Vancouver, Oregon
  - GSK Investigational Site, Abington, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, The Woodlands, Texas
- Austria (3):
  - GSK Investigational Site, Graz
  - GSK Investigational Site, Innsbruck
  - GSK Investigational Site, Vienna
- Belgium (4):
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Kortrijk
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
- Canada (6):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- Denmark (4):
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, Copenhagen
  - GSK Investigational Site, Herlev
  - GSK Investigational Site, Odense
- France (6):
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Saint-Brieuc
  - GSK Investigational Site, Saint-Herblain
- Germany (10):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Göttingen, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- GSK Investigational Site, Szolnok, Hungary
- Israel (7):
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Holon
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Rehovot
  - GSK Investigational Site, Tel Aviv
  - GSK Investigational Site, Tel Litwinsky
- Italy (5):
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Brescia, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Catania, Sicily
  - GSK Investigational Site, Milan
- Norway (2):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Oslo
- Poland (4):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Poznan
- Spain (4):
  - GSK Investigational Site, Oviedo, Principality of Asturias
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Palma de Mallorca
- Sweden (3):
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Stockholm
- United Kingdom (8):
  - GSK Investigational Site, Nottingham, Nottinghamshire
  - GSK Investigational Site, Yeovil, Somerset
  - GSK Investigational Site, Birmingham, West Midlands
  - GSK Investigational Site, Bebington, Wirral
  - GSK Investigational Site, London
  - GSK Investigational Site, Maidstone
  - GSK Investigational Site, Rhyl
  - GSK Investigational Site, Taunton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mirza MR, Monk BJ, Herrstedt J, Oza AM, Mahner S, Redondo A, Fabbro M, Ledermann JA, Lorusso D, Vergote I, Ben-Baruch NE, Marth C, Madry R, Christensen RD, Berek JS, Dorum A, Tinker AV, du Bois A, Gonzalez-Martin A, Follana P, Benigno B, Rosenberg P, Gilbert L, Rimel BJ, Buscema J, Balser JP, Agarwal S, Matulonis UA; ENGOT-OV16/NOVA Investigators. Niraparib Maintenance Therapy in Platinum-Sensitive, Recurrent Ovarian Cancer. N Engl J Med. 2016 Dec 1;375(22):2154-2164. doi: 10.1056/NEJMoa1611310. Epub 2016 Oct 7. PMID 27717299
- [Background] Mirza MR, Lindahl G, Mahner S, Redondo A, Fabbro M, Rimel BJ, Herrstedt J, Oza AM, Canzler U, Berek JS, Gonzalez-Martin A, Follana P, Lord R, Azodi M, Estenson K, Wang Z, Li Y, Gupta D, Matulonis U, Feng B. Ad hoc Analysis of the Phase III ENGOT-OV16/NOVA Study: Niraparib Efficacy in Germline BRCA Wild-type Recurrent Ovarian Cancer with Homologous Recombination Repair Defects. Cancer Res Commun. 2022 Nov 15;2(11):1436-1444. doi: 10.1158/2767-9764.CRC-22-0240. eCollection 2022 Nov. PMID 36970052
- [Derived] Monk BJ, Romero I, Graybill W, Churruca C, O'Malley DM, Knudsen AO, Yap OWS, Baurain JF, Rose PG, Denys H, Ghamande S, Pisano C, Fabbro M, Braicu EI, Calvert PM, Amit A, Prendergast E, Taylor A, Kheibarshekan L, Zhang ZY, Zajic S, Jewell RC, Gupta D, Gonzalez-Martin A. Niraparib Population Pharmacokinetics and Exposure-Response Relationships in Patients With Newly Diagnosed Advanced Ovarian Cancer. Clin Ther. 2024 Aug;46(8):612-621. doi: 10.1016/j.clinthera.2024.06.001. Epub 2024 Jul 16. PMID 39019698
- [Derived] Tattersall A, Ryan N, Wiggans AJ, Rogozinska E, Morrison J. Poly(ADP-ribose) polymerase (PARP) inhibitors for the treatment of ovarian cancer. Cochrane Database Syst Rev. 2022 Feb 16;2(2):CD007929. doi: 10.1002/14651858.CD007929.pub4. PMID 35170751
- [Derived] Mirza MR, Benigno B, Dorum A, Mahner S, Bessette P, Barcelo IB, Berton-Rigaud D, Ledermann JA, Rimel BJ, Herrstedt J, Lau S, du Bois A, Herraez AC, Kalbacher E, Buscema J, Lorusso D, Vergote I, Levy T, Wang P, de Jong FA, Gupta D, Matulonis UA. Long-term safety in patients with recurrent ovarian cancer treated with niraparib versus placebo: Results from the phase III ENGOT-OV16/NOVA trial. Gynecol Oncol. 2020 Nov;159(2):442-448. doi: 10.1016/j.ygyno.2020.09.006. Epub 2020 Sep 25. PMID 32981695
- [Derived] Matulonis UA, Walder L, Nottrup TJ, Bessette P, Mahner S, Gil-Martin M, Kalbacher E, Ledermann JA, Wenham RM, Woie K, Lau S, Marme F, Casado Herraez A, Hardy-Bessard AC, Banerjee S, Lindahl G, Benigno B, Buscema J, Travers K, Guy H, Mirza MR. Niraparib Maintenance Treatment Improves Time Without Symptoms or Toxicity (TWiST) Versus Routine Surveillance in Recurrent Ovarian Cancer: A TWiST Analysis of the ENGOT-OV16/NOVA Trial. J Clin Oncol. 2019 Dec 1;37(34):3183-3191. doi: 10.1200/JCO.19.00917. Epub 2019 Sep 16. PMID 31518175
- [Derived] Del Campo JM, Matulonis UA, Malander S, Provencher D, Mahner S, Follana P, Waters J, Berek JS, Woie K, Oza AM, Canzler U, Gil-Martin M, Lesoin A, Monk BJ, Lund B, Gilbert L, Wenham RM, Benigno B, Arora S, Hazard SJ, Mirza MR. Niraparib Maintenance Therapy in Patients With Recurrent Ovarian Cancer After a Partial Response to the Last Platinum-Based Chemotherapy in the ENGOT-OV16/NOVA Trial. J Clin Oncol. 2019 Nov 10;37(32):2968-2973. doi: 10.1200/JCO.18.02238. Epub 2019 Jun 7. PMID 31173551
- [Derived] Oza AM, Matulonis UA, Malander S, Hudgens S, Sehouli J, Del Campo JM, Berton-Rigaud D, Banerjee S, Scambia G, Berek JS, Lund B, Tinker AV, Hilpert F, Vazquez IP, D'Hondt V, Benigno B, Provencher D, Buscema J, Agarwal S, Mirza MR. Quality of life in patients with recurrent ovarian cancer treated with niraparib versus placebo (ENGOT-OV16/NOVA): results from a double-blind, phase 3, randomised controlled trial. Lancet Oncol. 2018 Aug;19(8):1117-1125. doi: 10.1016/S1470-2045(18)30333-4. Epub 2018 Jul 17. PMID 30026000
- [Derived] Berek JS, Matulonis UA, Peen U, Ghatage P, Mahner S, Redondo A, Lesoin A, Colombo N, Vergote I, Rosengarten O, Ledermann J, Pineda M, Ellard S, Sehouli J, Gonzalez-Martin A, Berton-Rigaud D, Madry R, Reinthaller A, Hazard S, Guo W, Mirza MR. Safety and dose modification for patients receiving niraparib. Ann Oncol. 2018 Aug 1;29(8):1784-1792. doi: 10.1093/annonc/mdy181. PMID 29767688
- See also: Facing our risk of cancer empowered website — http://www.facingourrisk.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, double-blind study conducted to analyze maintenance with niraparib versus placebo in participants with ovarian cancer.
Pre-assignment Details: A total of 596 participants were enrolled in the study. The results presented are based on the data cut-off date of 31 March 2021 (which aligns with the time of the study unblinding) and the post-unblinding safety data until the end of study (01-April-2021 to 26-December-2021).
Groups:
- gBRCA Niraparib: Participants with germline breast cancer gene (gBRCA) mutation received oral dose of niraparib 300 milligrams (mg) once daily in 28-day cycles until disease progression.
- gBRCA Placebo: Participants with germline BRCA mutation received oral dose of placebo matching niraparib once daily in 28-day cycles until disease progression.
- Non-gBRCA Niraparib: Participants without germline BRCA mutation received oral dose of niraparib 300 mg once daily orally in 28-day cycles until disease progression.
- Non-gBRCA Placebo: Participants without germline BRCA mutation received matching placebo once daily orally in 28-day cycles until disease progression
- FE Sub-study: Fasted/Fed: Participants received a single dose of 3x100 mg capsules of niraparib administered orally following a minimum 10-hour overnight fast in Period 1 followed by 300 mg capsules of niraparib administered orally as single dose in fed condition (high-fat meal) in Period 2. There was a washout period of 7 days between treatment periods.
- FE Sub-study: Fed/Fasted: Participants received single dose of 3x100 mg capsules of niraparib administered orally following a high-fat meal in Period 1 followed by 3x100 mg capsules of niraparib administered orally as single dose in fasted condition in Period 2. There was a washout period of 7 days between treatment periods.
- QTc Sub-study: Niraparib: Participants received Niraparib 300 mg once daily orally.
- gBRCA Niraparib (Post-study Unblinding [PSU]): Participants with germline breast cancer gene (gBRCA) mutation received oral dose of niraparib 300 milligrams (mg) once daily in 28-day cycles until disease progression. This arm presents data for post-study unblinding duration 01-Apr-2021 to 26-Dec-2021
- gBRCA Placebo (PSU): Participants with germline BRCA mutation received oral dose of placebo matching niraparib once daily in 28-day cycles until disease progression. This arm presents data for post-study unblinding duration 01-Apr-2021 to 26-Dec-2021
- Non-gBRCA Niraparib (PSU): Participants without germline BRCA mutation received oral dose of niraparib 300 mg once daily orally in 28-day cycles until disease progression. This arm presents data for post-study unblinding duration 01-Apr-2021 to 26-Dec-2021
- Non-gBRCA Placebo (PSU): Participants without germline BRCA mutation received matching placebo once daily orally in 28-day cycles until disease progression. This arm presents data for post-study unblinding duration 01-Apr-2021 to 26-Dec-2021
Period: Main Study (Upto 7years 7months 6 Days)
Arm/Group | gBRCA Niraparib | gBRCA Placebo | Non-gBRCA Niraparib | Non-gBRCA Placebo | FE Sub-study: Fasted/Fed | FE Sub-study: Fed/Fasted | QTc Sub-study: Niraparib | gBRCA Niraparib (Post-study Unblinding [PSU]) | gBRCA Placebo (PSU) | Non-gBRCA Niraparib (PSU) | Non-gBRCA Placebo (PSU)
Started | 138 | 65 | 234 | 116 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 138 | 65 | 234 | 116 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Ongoing at the time of analysis | 22 | 8 | 31 | 13 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 20 | 11 | 29 | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 7 | 2 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disease progression | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Subject unblinded by sponsor | 12 | 12 | 15 | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 72 | 29 | 146 | 68 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other reasons | 5 | 3 | 8 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: FE Sub-study, Period1 (Day1)
Arm/Group | gBRCA Niraparib | gBRCA Placebo | Non-gBRCA Niraparib | Non-gBRCA Placebo | FE Sub-study: Fasted/Fed | FE Sub-study: Fed/Fasted | QTc Sub-study: Niraparib | gBRCA Niraparib (Post-study Unblinding [PSU]) | gBRCA Placebo (PSU) | Non-gBRCA Niraparib (PSU) | Non-gBRCA Placebo (PSU)
Started | 0 | 0 | 0 | 0 | 8 | 9 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 8 | 8 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: FE Sub-study, Washout 1 (Up to Day 7)
Arm/Group | gBRCA Niraparib | gBRCA Placebo | Non-gBRCA Niraparib | Non-gBRCA Placebo | FE Sub-study: Fasted/Fed | FE Sub-study: Fed/Fasted | QTc Sub-study: Niraparib | gBRCA Niraparib (Post-study Unblinding [PSU]) | gBRCA Placebo (PSU) | Non-gBRCA Niraparib (PSU) | Non-gBRCA Placebo (PSU)
Started | 0 | 0 | 0 | 0 | 8 | 8 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 7 | 8 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Transferred to Other Arm/Group | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: FE Sub-study, Period 2 (Day 1)
Arm/Group | gBRCA Niraparib | gBRCA Placebo | Non-gBRCA Niraparib | Non-gBRCA Placebo | FE Sub-study: Fasted/Fed | FE Sub-study: Fed/Fasted | QTc Sub-study: Niraparib | gBRCA Niraparib (Post-study Unblinding [PSU]) | gBRCA Placebo (PSU) | Non-gBRCA Niraparib (PSU) | Non-gBRCA Placebo (PSU)
Started | 0 | 0 | 0 | 0 | 7 | 8 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 7 | 8 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: QTcSub-study(Upto 5 Year,10 Month,22day)
Arm/Group | gBRCA Niraparib | gBRCA Placebo | Non-gBRCA Niraparib | Non-gBRCA Placebo | FE Sub-study: Fasted/Fed | FE Sub-study: Fed/Fasted | QTc Sub-study: Niraparib | gBRCA Niraparib (Post-study Unblinding [PSU]) | gBRCA Placebo (PSU) | Non-gBRCA Niraparib (PSU) | Non-gBRCA Placebo (PSU)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0
Not completed — Other Reasons | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0 | 0 | 0 | 0
Period: Main Study PSU (Up to 8months, 26days)
Arm/Group | gBRCA Niraparib | gBRCA Placebo | Non-gBRCA Niraparib | Non-gBRCA Placebo | FE Sub-study: Fasted/Fed | FE Sub-study: Fed/Fasted | QTc Sub-study: Niraparib | gBRCA Niraparib (Post-study Unblinding [PSU]) | gBRCA Placebo (PSU) | Non-gBRCA Niraparib (PSU) | Non-gBRCA Placebo (PSU)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 22 | 8 | 31 | 13
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 22 | 8 | 31 | 13
Not completed — Subject Unblinded by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 8 | 18 | 12
Not completed — Subject Moved to Rollover Study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 9 | 0
Not completed — Other reasons | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population was the intent-to-treat population, defined as all randomized participants with participants analyzed according to the study drug assigned via randomization
Groups:
- Total: Total of all reporting groups
Arm/Group | gBRCA Niraparib | gBRCA Placebo | Non-gBRCA Niraparib | Non-gBRCA Placebo | FE Sub-study: Fasted/Fed | FE Sub-study: Fed/Fasted | QTc Sub-study: Niraparib | Total
Number analyzed (Participants) | 138 | 65 | 234 | 116 | 8 | 9 | 26 | 596
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 64 years | 110 | 49 | 130 | 69 | 5 | 5 | 16 | 384
  >=65 years | 28 | 16 | 104 | 47 | 3 | 4 | 10 | 212
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 65 | 234 | 116 | 8 | 9 | 26 | 596
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Asian | 2 | 3 | 10 | 4 | 0 | 0 | 1 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 1 | 1 | 4 | 1 | 1 | 0 | 3 | 11
  White | 123 | 55 | 201 | 101 | 6 | 9 | 21 | 516
  Unknown or Not Reported | 11 | 6 | 19 | 10 | 0 | 0 | 0 | 46

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) in Cohort With Germline BReast CAncer Gene (BRCA) Mutation (gBRCA)
Description: PFS was defined as the time between randomization and disease progression or death from any cause. Computed tomography or magnetic resonance imaging to assess disease progression was performed at baseline, every 8 weeks through cycle 14, and then every 12 weeks until treatment discontinuation. The objective assessment of disease progression was determined by means of central radiologic and clinical review, according to Response Evaluation Criteria in Solid Tumors (RECIST),version 1.1, which was performed in a blinded fashion. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: From date of randomization to the earliest date of disease progression or death from any cause, up to 7 years 7 months and 4 days
Population: Intent-to-treat population was defined as all randomized participants with participants analyzed according to the study drug assigned via randomization
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | gBRCA Niraparib | gBRCA Placebo
Number analyzed (Participants) | 138 | 65
months | 21 [12.9 to NA] — Upper limit of confidence interval (CI) was not estimable as upper limits of CI for survivor function were above 0.5 (SAS PROC LIFETEST). | 5.5 [3.8 to 7.2]
Statistical Analysis 1: Comparison: gBRCA Niraparib vs gBRCA Placebo; Test type: Superiority; p < 0.0001, Log Rank — Two-sided P-value. PFS was independently evaluated in gBRCAmut cohort and non-gBRCAmut cohort; Strata: tm to progression after penultimate platinum tx; use of bevacizumab w/penultimate or last platinum tx; best response during last platinum tx; Hazard Ratio (HR) = 0.27, 95% CI 2-sided [0.173 to 0.410] — Niraparib:Placebo, based on the stratified Cox Proportional Hazards Model using randomization stratification factors

2. Primary Outcome: Progression-Free Survival (PFS) in Cohort With No Germline BCRA With Homologous Recombination Deficiency-positive (HRD+) Tumors (Non-gBRCAmut HRD+)
Description: PFS was defined as the time between randomization and disease progression or death from any cause. Computed tomography or magnetic resonance imaging to assess disease progression was performed at baseline, every 8 weeks through cycle 14, and then every 12 weeks until treatment discontinuation. The objective assessment of disease progression was determined by means of central radiologic and clinical review, according to Response Evaluation Criteria in Solid Tumors (RECIST),version 1.1, which was performed in a blinded fashion. PD was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: From date of randomization to the earliest date of disease progression or death from any cause, up to 7 years, 7 months and 4 days
Population: Intent-to-treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Non-gBRCAmut HRD+ Niraparib: Niraparib (300 mg) once daily in 28-day cycles until disease progression in participants with homologous recombination deficiency-positive (HRD+) tumors Niraparib vs. Placebo 2:1 ratio
- Non-gBRCAmut HRD+ Placebo: Placebo once daily in 28-day cycles until disease progression patients with homologous recombination deficiency-positive (HRD+) tumors Niraparib vs. Placebo 2:1 ratio
Arm/Group | Non-gBRCAmut HRD+ Niraparib | Non-gBRCAmut HRD+ Placebo
Number analyzed (Participants) | 106 | 56
months | 12.9 [8.1 to 15.9] | 3.8 [3.5 to 5.7]
Statistical Analysis 1: Comparison: Non-gBRCAmut HRD+ Niraparib vs Non-gBRCAmut HRD+ Placebo; Test type: Superiority; p < 0.0001, Log Rank — Two-sided P-value. PFS was independently evaluated in gBRCAmut cohort and non-gBRCAmut cohort. Hierarchical testing: HRD+ subset tested first. If HRD+ subset demonstrated statistical significance, overall non-gBRCA cohort was then tested; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.38, 95% CI 2-sided [0.243 to 0.586] — Niraparib:Placebo, based on the stratified Cox Proportional Hazards Model using randomization stratification factors

3. Primary Outcome: Progression-Free Survival (PFS) in Cohort With No Germline BRCA Mutation
Description: PFS was defined as the time between randomization and disease progression or death from any cause. Computed tomography or magnetic resonance imaging to assess disease progression was performed at baseline, every 8 weeks through cycle 14, and then every 12 weeks until treatment discontinuation. The objective assessment of disease progression was determined by means of central radiologic and clinical review, according to Response Evaluation Criteria in Solid Tumors (RECIST),version 1.1, which was performed in a blinded fashion.PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: as for outcome 2
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Non-gBRCA Niraparib: Niraparib (300 mg) once daily in 28-day cycles until disease progression in patients without germline BRCA mutation Niraparib vs. Placebo 2:1 ratio
- Non-gBRCA Placebo: Placebo once daily in 28-day cycles until disease progression in patients without germline BRCA mutation Niraparib vs. Placebo 2:1 ratio
Arm/Group | Non-gBRCA Niraparib | Non-gBRCA Placebo
Number analyzed (Participants) | 234 | 116
Months | 9.3 [7.2 to 11.2] | 3.9 [3.7 to 5.5]
Statistical Analysis 1: Comparison: Non-gBRCA Niraparib vs Non-gBRCA Placebo; Test type: Superiority; p < 0.0001, Log Rank — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.338 to 0.607] — Niraparib:Placebo, based on the stratified Cox Proportional Hazards Model using randomization stratification factors

4. Secondary Outcome: Time to First Subsequent Therapy in Cohort With Germline BRCA Mutation (gBRCA)
Description: The TFST was defined as the time from the date of randomization to the start date of the first subsequent anti-cancer therapy or death.
Time Frame: From date of randomization to the earliest date of first subsequent therapy or death, up to 7 years, 7 months and 4 days
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | gBRCA Niraparib | gBRCA Placebo
Number analyzed (Participants) | 138 | 65
Months | 19.1 [14.6 to 21.9] | 8.6 [6.9 to 12.2]
Statistical Analysis 1: Comparison: gBRCA Niraparib vs gBRCA Placebo; Test type: Superiority; p = 0.0005, Log Rank — Two-sided p-value; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.412 to 0.783]

5. Secondary Outcome: Time to First Subsequent Therapy in Cohort With No Germline BRCA Mutation
Description: as for outcome 4
Time Frame: as for outcome 4
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Non-gBRCA Niraparib | Non-gBRCA Placebo
Number analyzed (Participants) | 234 | 116
Months | 12.4 [10.9 to 14.5] | 7.4 [5.9 to 8.7]
Statistical Analysis 1: Comparison: Non-gBRCA Niraparib vs Non-gBRCA Placebo; Test type: Superiority; p < 0.0001, Log Rank — Two-sided P-value; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.454 to 0.740]

6. Secondary Outcome: Chemotherapy-Free Interval in Cohort With Germline BRCA Mutation (gBRCA)
Description: Chemotherapy-Free Interval was defined as the time from the last platinum therapy prior to randomization to the initiation of the next anti-cancer therapy after maintenance treatment
Time Frame: From date of last platinum therapy prior to randomization to the initiation of the next anti-cancer therapy after maintenance treatment, up to 7 years, 7 months and 4 days
Population: Intent-to-treat Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | gBRCA Niraparib | gBRCA Placebo
Number analyzed (Participants) | 138 | 65
Months | 20.0 [16.2 to 23.3] | 9.4 [7.9 to 10.4]
Statistical Analysis 1: Comparison: gBRCA Niraparib vs gBRCA Placebo; Test type: Superiority; p < 0.0001, Log Rank — Two-sided P-value; Hazard Ratio (HR) = 0.39, 95% CI 2-sided [0.268 to 0.561]

7. Secondary Outcome: Chemotherapy-Free Interval in Cohort With No Germline BRCA Mutation
Description: as for outcome 6
Time Frame: as for outcome 6
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Non-gBRCA Niraparib | Non-gBRCA Placebo
Number analyzed (Participants) | 234 | 116
Months | 13.4 [11.3 to 14.8] | 8.7 [6.9 to 10.0]
Statistical Analysis 1: Comparison: Non-gBRCA Niraparib vs Non-gBRCA Placebo; Test type: Superiority; p < 0.0001, Log Rank — Two-sided P-value; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.428 to 0.727]

8. Secondary Outcome: Progression-Free Survival 2 in Cohort With Germline BRCA Mutation (gBRCA)
Description: Progression-Free Survival 2 was defined as the date of randomization in the current study to the earlier date of assessment of progression on the next anti-cancer therapy following study treatment or death due to any cause. Progression was determined by the investigator via clinical and radiographic assessment using the same criteria as used in the current study.
Time Frame: From treatment randomization to the earlier of the date of disease progression on the next anti-cancer therapy following study treatment or death due to any cause, up to 7 years, 7 months and 4 days
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | gBRCA Niraparib | gBRCA Placebo
Number analyzed (Participants) | 138 | 65
Months | 29.9 [24.8 to 33.4] | 22.7 [19.5 to 25.9]
Statistical Analysis 1: Comparison: gBRCA Niraparib vs gBRCA Placebo; Test type: Superiority; p = 0.0302, Log Rank — Two-sided P-value; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.500 to 0.968]

9. Secondary Outcome: Progression-Free Survival 2 in Cohort With No Germline BRCA Mutation
Description: as for outcome 8
Time Frame: as for outcome 8
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Non-gBRCA Niraparib | Non-gBRCA Placebo
Number analyzed (Participants) | 234 | 116
Months | 19.5 [17.1 to 22.3] | 16.1 [13.6 to 22.8]
Statistical Analysis 1: Comparison: Non-gBRCA Niraparib vs Non-gBRCA Placebo; Test type: Superiority; p = 0.0748, Log Rank — Two-sided P-value; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.627 to 1.022]

10. Secondary Outcome: Overall Survival in Cohort With Germline BRCA Mutation (gBRCA)
Description: Overall survival was defined as the date of randomization to the date of death by any cause.
Time Frame: From treatment randomization to date of death by any cause, up to 7 years, 7 months and 4 days
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | gBRCA Niraparib | gBRCA Placebo
Number analyzed (Participants) | 138 | 65
Months | 40.9 [34.9 to 52.9] | 38.1 [27.6 to 47.3]
Statistical Analysis 1: Comparison: gBRCA Niraparib vs gBRCA Placebo; Test type: Superiority; p = 0.3580, Log Rank — Two-sided P-value; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.606 to 1.198]

11. Secondary Outcome: Overall Survival in Cohort With No Germline BRCA Mutation
Description: Overall survival was defined as the date of randomization to the date of death by any cause.
Time Frame: From treatment randomization to date of death by any cause, up to 7 years, 7 months and 4 days
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Non-gBRCA Niraparib | Non-gBRCA Placebo
Number analyzed (Participants) | 234 | 116
Months | 31.0 [27.8 to 35.6] | 34.8 [27.9 to 41.4]
Statistical Analysis 1: Comparison: Non-gBRCA Niraparib vs Non-gBRCA Placebo; Test type: Superiority; p = 0.6868, Log Rank — Two-sided P-value; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.813 to 1.369]

12. Secondary Outcome: Time to Second Subsequent Therapy in Cohort With Germline BRCA Mutation (gBRCA)
Description: TSST was defined as the date of randomization to the earlier of the start date of second follow-up anti-cancer treatment or death.
Time Frame: From the date of randomization to the start date of the second subsequent anti-cancer therapy, up to 7 years, 7 months and 4 days
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | gBRCA Niraparib | gBRCA Placebo
Number analyzed (Participants) | 138 | 65
Months | 29.7 [23.3 to 33.4] | 19.6 [14.4 to 25.5]
Statistical Analysis 1: Comparison: gBRCA Niraparib vs gBRCA Placebo; Test type: Superiority; p = 0.0061, Log Rank — Two-sided P-value; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.451 to 0.878]

13. Secondary Outcome: Time to Second Subsequent Therapy in Cohort With No Germline BRCA Mutation
Description: as for outcome 12
Time Frame: as for outcome 12
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Non-gBRCA Niraparib | Non-gBRCA Placebo
Number analyzed (Participants) | 234 | 116
Months | 20.3 [18.0 to 23.4] | 16.7 [14.9 to 21.3]
Statistical Analysis 1: Comparison: Non-gBRCA Niraparib vs Non-gBRCA Placebo; Test type: Superiority; p = 0.1674, Log Rank — Two-sided P-value; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.654 to 1.077]

14. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Ovarian Symptom Index in Cohort With Germline BRCA at Cycle 2
Description: Functional Assessment of Cancer Therapy-Ovarian Symptom Index is a validated, 8-item measure of symptom response to treatment for ovarian cancer. Participants respond to their symptom experience over the past 7 days using a 5-point Likert scale score from "not at all" (0) to "very much" (4). The total score was calculated by multiplying the sum of all items scored by 8 and dividing the result by the number of responses. The total symptom index was calculated as the total of the 8 scores, ranging from 0 ("severely symptomatic") to 32 ("asymptomatic"). A positive change from Baseline indicates improvement. Baseline was latest non-missing pre-dose assessment on or before randomization date. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (pre-dose on Day 1) and at Cycle 2 (Each cycle was of 28 days)
Population: Intent-to-treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | gBRCA Niraparib | gBRCA Placebo
Number analyzed (Participants) | 114 | 55
Scores on a scale | -0.8 (4.58) | -0.3 (3.19)

15. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Ovarian Symptom Index in Cohort With Germline BRCA at Cycle 4
Description: as for outcome 14
Time Frame: Baseline (Pre-dose on Day 1) and at Cycle 4 (Each cycle was of 28 days)
Population: Intent-to-treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | gBRCA Niraparib | gBRCA Placebo
Number analyzed (Participants) | 109 | 43
Scores on a scale | -0.1 (4.07) | -0.3 (3.88)

16. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Ovarian Symptom Index in Cohort With Germline BRCA at Cycle 6
Description: as for outcome 14
Time Frame: Baseline (pre-dose on Day 1) and at Cycle 6 (Each cycle was of 28 days)
Population: Intent-to-treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | gBRCA Niraparib | gBRCA Placebo
Number analyzed (Participants) | 95 | 36
Scores on a scale | 0.5 (3.77) | -0.5 (4.27)

17. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Ovarian Symptom Index in Cohort With Germline BRCA at Post-progression
Description: as for outcome 14
Time Frame: Baseline (Pre-dose on Cycle 1 Day 1, Each cycle was of 28 days) and up to 7 years, 7 months and 4 days
Population: Intent-to-treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | gBRCA Niraparib | gBRCA Placebo
Number analyzed (Participants) | 80 | 37
Scores on a scale | -0.751 (4.4342) | -1.324 (4.5034)

18. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Ovarian Symptom Index in Cohort With no Germline BRCA at Cycle 2
Description: as for outcome 14
Time Frame: Baseline (Pre-dose on Day 1) and at Cycle 2 (Each cycle was of 28 days)
Population: Intent-to-treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Non-gBRCA Niraparib | Non-gBRCA Placebo
Number analyzed (Participants) | 181 | 97
Scores on a scale | -1.0 (3.79) | -0.3 (2.84)

19. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Ovarian Symptom Index in Cohort With no Germline BRCA at Cycle 4
Description: as for outcome 14
Time Frame: Baseline (Pre-dose on Day 1) and at Cycle 4 (Each cycle was of 28 days)
Population: Intent-to-treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Non-gBRCA Niraparib | Non-gBRCA Placebo
Number analyzed (Participants) | 150 | 77
Scores on a scale | -0.7 (4.16) | -0.9 (4.23)

20. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Ovarian Symptom Index in Cohort With no Germline BRCA at Cycle 6
Description: as for outcome 14
Time Frame: Baseline (Pre-dose on Day 1) and at Cycle 6 (Each cycle was of 28 days)
Population: Intent-to-treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Non-gBRCA Niraparib | Non-gBRCA Placebo
Number analyzed (Participants) | 124 | 50
Scores on a scale | -0.2 (3.76) | -0.9 (3.43)

21. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Ovarian Symptom Index in Cohort With no Germline BRCA at Post-progression
Description: as for outcome 14
Time Frame: Baseline (Pre-dose on Day 1) and up to 7 years, 7 months and 4 days
Population: Intent-to-treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Non-gBRCA Niraparib | Non-gBRCA Placebo
Number analyzed (Participants) | 146 | 82
Scores on a scale | -2.595 (5.5700) | -1.801 (4.0290)

22. Secondary Outcome: Change From Baseline in European Quality of Life Scale, 5-Dimensions (EQ-5D-5L) in Cohort With Germline BRCA at Cycle 2
Description: EQ-5D-5L is a well-validated, general preference-based, health-related Quality of Life (QoL) instrument. The EQ-5D-5L encompasses 5 domains, asking participants to rate their perceived health state today on the following dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each domain has 5 possible levels: "no problems" (Level 1), "slight problems" (Level 2), "moderate problems" (Level 3), "severe problems" (Level 4), and "extreme problems" (Level 5). Responses for 5 dimensions together formed a 5-figure description of health state (e.g.11111 indicates no problems in all 5 dimensions). Baseline was latest non-missing pre-dose assessment on or before randomization date. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Pre-dose on Day 1) and at Cycle 2 (Each cycle was of 28 days)
Population: Intent-to-treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | gBRCA Niraparib | gBRCA Placebo
Number analyzed (Participants) | 118 | 59
Scores on a scale | -0.008 (0.1092) | -0.008 (0.1354)

23. Secondary Outcome: Change From Baseline in EQ-5D-5L in Cohort With Germline BRCA at Cycle 4
Description: as for outcome 22
Time Frame: Baseline (Pre-dose on Day 1) and at Cycle 4 (Each cycle was of 28 days)
Population: Intent-to-treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | gBRCA Niraparib | gBRCA Placebo
Number analyzed (Participants) | 113 | 44
Scores on a scale | -0.010 (0.1225) | -0.035 (0.1156)

24. Secondary Outcome: Change From Baseline in EQ-5D-5L in Cohort With Germline BRCA at Cycle 6
Description: as for outcome 22
Time Frame: Baseline (Pre-dose on Day 1) and at Cycle 6 (Each cycle was of 28 days)
Population: Intent-to-treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | gBRCA Niraparib | gBRCA Placebo
Number analyzed (Participants) | 99 | 36
Scores on a scale | 0.002 (0.1116) | -0.004 (0.1463)

25. Secondary Outcome: Change From Baseline in EQ-5D-5L in Cohort With Germline BRCA at Post-progression
Description: as for outcome 22
Time Frame: Baseline (Pre-dose on Day 1) and up to 7 years, 7 months and 4 days
Population: Intent-to-treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | gBRCA Niraparib | gBRCA Placebo
Number analyzed (Participants) | 81 | 38
Scores on a scale | -0.041 (0.1192) | -0.013 (0.1580)

26. Secondary Outcome: Change From Baseline in EQ-5D-5L in Cohort With no Germline BRCA at Cycle 2
Description: as for outcome 22
Time Frame: Baseline (Pre-dose on Day 1) and at Cycle 2 (Each cycle was of 28 days)
Population: Intent-to-treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Non-gBRCA Niraparib | Non-gBRCA Placebo
Number analyzed (Participants) | 185 | 96
Scores on a scale | -0.007 (0.1013) | -0.011 (0.1015)

27. Secondary Outcome: Change From Baseline in EQ-5D-5L in Cohort With no Germline BRCA at Cycle 4
Description: as for outcome 22
Time Frame: Baseline (Pre-dose on Day 1) and at Cycle 4 (Each cycle was of 28 days)
Population: Intent-to-treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Non-gBRCA Niraparib | Non-gBRCA Placebo
Number analyzed (Participants) | 155 | 80
Scores on a scale | -0.004 (0.1077) | -0.014 (0.0870)

28. Secondary Outcome: Change From Baseline in EQ-5D-5L in Cohort With no Germline BRCA at Cycle 6
Description: as for outcome 22
Time Frame: Baseline (Pre-dose on Day 1) and at Cycle 6 (Each cycle was of 28 days)
Population: Intent-to-treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Non-gBRCA Niraparib | Non-gBRCA Placebo
Number analyzed (Participants) | 127 | 50
Scores on a scale | 0.005 (0.1097) | -0.011 (0.0949)

29. Secondary Outcome: Change From Baseline in EQ-5D-5L in Cohort With no Germline BRCA at Post-progression
Description: as for outcome 22
Time Frame: Baseline (Pre-dose on Day 1) and up to 7 years, 7 months and 4 days
Population: Intent-to-treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Non-gBRCA Niraparib | Non-gBRCA Placebo
Number analyzed (Participants) | 149 | 84
Scores on a scale | -0.047 (0.1355) | -0.050 (0.1351)

30. Secondary Outcome: Number of Participants With Response to Neuropathy Questionnaire in Cohort With Germline BRCA at Baseline
Description: A Neuropathy Questionnaire measures the participant's symptom experience over the past 7 days using a 5-point Likert scale of "not at all" (0) to "very much" (4). There are 2 items that ask if the participant's feet (item 1) or hands (item 2) feel numb or have prickling/tingling feelings. The Neuropathy Questionnaire was used to determine the chemotherapy-induced peripheral neuropathy (CIPN) status of each participant as well as provide an anchor for interpreting the impact of CIPN on participant's QoL. Two thresholds were used. For the first, a participant was determined to have CIPN if a score greater than 0 ("not at all") was recorded for either item. For the second, CIPN was assigned if a participant recorded a score greater than 1 ("a little bit"). Baseline was latest non-missing pre-dose assessment on or before randomization date.
Time Frame: At Baseline
Population: Intent-to-treat Population.
Measure: Count of Participants; unit: Participants
Arm/Group | gBRCA Niraparib | gBRCA Placebo
Number analyzed (Participants) | 138 | 65
Participants
  Feet, 0-Not at all | 47 | 26
  Feet, 1-A little bit | 32 | 12
  Feet, 2-Somewhat | 24 | 9
  Feet, 3-Quite a bit | 21 | 10
  Feet, 4-Very much | 9 | 6
  Hands, 0-Not at all | 80 | 37
  Hands, 1-A little bit | 28 | 13
  Hands, 2-Somewhat | 8 | 6
  Hands, 3-Quite a bit | 14 | 5
  Hands, 4-Very much | 3 | 2
Statistical Analysis 1: Comparison: gBRCA Niraparib vs gBRCA Placebo; Test type: Superiority; p = 0.7969, Pearson's Chi-squared test; Analysis for gBRCA Niraparib vs gBRCA Placebo-Feet
Statistical Analysis 2: Comparison: gBRCA Niraparib vs gBRCA Placebo; Test type: Superiority; p = 0.8794, Pearson's Chi-squared test; Analysis for gBRCA Niraparib vs gBRCA Placebo-Hands

31. Secondary Outcome: Number of Participants With Response to Neuropathy Questionnaire in Cohort With Germline BRCA at Cycle 2
Description: A Neuropathy Questionnaire measures the participant's symptom experience over the past 7 days using a 5-point Likert scale of "not at all" (0) to "very much" (4). There are 2 items that ask if the participant's feet (item 1) or hands (item 2) feel numb or have prickling/tingling feelings. The Neuropathy Questionnaire was used to determine the chemotherapy-induced peripheral neuropathy (CIPN) status of each participant as well as provide an anchor for interpreting the impact of CIPN on participant's QoL. Two thresholds were used. For the first, a participant was determined to have CIPN if a score greater than 0 ("not at all") was recorded for either item. For the second, CIPN was assigned if a participant recorded a score greater than 1 ("a little bit").
Time Frame: At Cycle 2 (Each cycle was of 28 days)
Population: Intent-to-treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | gBRCA Niraparib | gBRCA Placebo
Number analyzed (Participants) | 132 | 64
Participants
  Feet, 0-Not at all | 48 | 25
  Feet, 1-A little bit | 22 | 5
  Feet, 2-Somewhat | 17 | 15
  Feet, 3-Quite a bit | 20 | 10
  Feet, 4-Very much | 8 | 3
  Hands, 0-Not at all | 73 | 31
  Hands, 1-A little bit | 19 | 16
  Hands, 2-Somewhat | 13 | 6
  Hands, 3-Quite a bit | 7 | 2
  Hands, 4-Very much | 3 | 2
Statistical Analysis 1: Comparison: gBRCA Niraparib vs gBRCA Placebo; Test type: Superiority; p = 0.2399, Pearson's Chi-squared test; Analysis for gBRCA Niraparib vs gBRCA Placebo-Feet
Statistical Analysis 2: Comparison: gBRCA Niraparib vs gBRCA Placebo; Test type: Superiority; p = 0.4584, Pearson's Chi-squared test; Analysis for gBRCA Niraparib vs gBRCA Placebo-Hands

32. Secondary Outcome: Number of Participants With Response to Neuropathy Questionnaire in Cohort With Germline BRCA at Cycle 4
Description: as for outcome 31
Time Frame: At Cycle 4 (Each cycle was of 28 days)
Population: Intent-to-treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | gBRCA Niraparib | gBRCA Placebo
Number analyzed (Participants) | 120 | 54
Participants
  Feet, 0-Not at all | 47 | 20
  Feet, 1-A little bit | 22 | 6
  Feet, 2-Somewhat | 20 | 7
  Feet, 3-Quite a bit | 15 | 8
  Feet, 4-Very much | 6 | 2
  Hands, 0-Not at all | 70 | 29
  Hands, 1-A little bit | 18 | 6
  Hands, 2-Somewhat | 16 | 3
  Hands, 3-Quite a bit | 4 | 4
  Hands, 4-Very much | 2 | 1
Statistical Analysis 1: Comparison: gBRCA Niraparib vs gBRCA Placebo; Test type: Superiority; p = 0.8566, Pearson's Chi-squared test; Analysis for gBRCA Niraparib vs gBRCA Placebo-Feet
Statistical Analysis 2: Comparison: gBRCA Niraparib vs gBRCA Placebo; Test type: Superiority; p = 0.4705, Pearson's Chi-squared test; Analysis for gBRCA Niraparib vs gBRCA Placebo-Hands

33. Secondary Outcome: Number of Participants With Response to Neuropathy Questionnaire in Cohort With Germline BRCA at Cycle 6
Description: as for outcome 31
Time Frame: At Cycle 6 (Each cycle was of 28 days)
Population: Intent-to-treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | gBRCA Niraparib | gBRCA Placebo
Number analyzed (Participants) | 105 | 41
Participants
  Feet, 0-Not at all | 44 | 17
  Feet, 1-A little bit | 17 | 5
  Feet, 2-Somewhat | 13 | 7
  Feet, 3-Quite a bit | 15 | 5
  Feet, 4-Very much | 9 | 2
  Hands, 0-Not at all | 54 | 21
  Hands, 1-A little bit | 25 | 8
  Hands, 2-Somewhat | 10 | 4
  Hands, 3-Quite a bit | 6 | 2
  Hands, 4-Very much | 2 | 1
Statistical Analysis 1: Comparison: gBRCA Niraparib vs gBRCA Placebo; Test type: Superiority; p = 0.8521, Pearson's Chi-squared test; Analysis for gBRCA Niraparib vs gBRCA Placebo-Feet
Statistical Analysis 2: Comparison: gBRCA Niraparib vs gBRCA Placebo; Test type: Superiority; p = 0.9923, Pearson's Chi-squared test; Analysis for gBRCA Niraparib vs gBRCA Placebo-Hands

34. Secondary Outcome: Number of Participants With Response to Neuropathy Questionnaire in Cohort With Germline BRCA at Post-progression
Description: as for outcome 31
Time Frame: Up to 7 years, 7 months and 4 days
Population: Intent-to-treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | gBRCA Niraparib | gBRCA Placebo
Number analyzed (Participants) | 104 | 49
Participants
  Feet, 0-Not at all | 31 | 15
  Feet, 1-A little bit | 20 | 9
  Feet, 2-Somewhat | 7 | 3
  Feet, 3-Quite a bit | 15 | 7
  Feet, 4-Very much | 7 | 3
  Hands, 0-Not at all | 44 | 26
  Hands, 1-A little bit | 18 | 4
  Hands, 2-Somewhat | 8 | 3
  Hands, 3-Quite a bit | 7 | 4
  Hands, 4-Very much | 3 | 0
Statistical Analysis 1: Comparison: gBRCA Niraparib vs gBRCA Placebo; Test type: Superiority; p = 0.9997, Pearson's Chi-squared test; Analysis for gBRCA Niraparib vs gBRCA Placebo-Feet
Statistical Analysis 2: Comparison: gBRCA Niraparib vs gBRCA Placebo; Test type: Superiority; p = 0.3518, Pearson's Chi-squared test; Analysis for gBRCA Niraparib vs gBRCA Placebo-Hands

35. Secondary Outcome: Number of Participants With Response to Neuropathy Questionnaire in Cohort With no Germline BRCA at Baseline
Description: as for outcome 30
Time Frame: At Baseline
Population: Intent-to-treat Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-gBRCA Niraparib | Non-gBRCA Placebo
Number analyzed (Participants) | 234 | 116
Participants
  Feet, 0-Not at all | 71 | 40
  Feet, 1-A little bit | 58 | 26
  Feet, 2-Somewhat | 37 | 16
  Feet, 3-Quite a bit | 43 | 21
  Feet, 4-Very much | 18 | 9
  Hands, 0-Not at all | 120 | 48
  Hands, 1-A little bit | 56 | 37
  Hands, 2-Somewhat | 28 | 12
  Hands, 3-Quite a bit | 15 | 11
  Hands, 4-Very much | 8 | 2
Statistical Analysis 1: Comparison: Non-gBRCA Niraparib vs Non-gBRCA Placebo; Test type: Superiority; p = 0.9367, Pearson's Chi-squared test; Analysis for gBRCA Niraparib vs gBRCA Placebo-Hands
Statistical Analysis 2: Comparison: Non-gBRCA Niraparib vs Non-gBRCA Placebo; Test type: Superiority; p = 0.2502, Pearson's Chi-squared test; Analysis for gBRCA Niraparib vs gBRCA Placebo-Hands

36. Secondary Outcome: Number of Participants With Response to Neuropathy Questionnaire in Cohort With no Germline BRCA at Cycle 2
Description: as for outcome 31
Time Frame: At Cycle 2 (Each cycle was of 28 days)
Population: Intent-to-treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-gBRCA Niraparib | Non-gBRCA Placebo
Number analyzed (Participants) | 212 | 113
Participants
  Feet, 0-Not at all | 69 | 32
  Feet, 1-A little bit | 39 | 17
  Feet, 2-Somewhat | 30 | 12
  Feet, 3-Quite a bit | 34 | 18
  Feet, 4-Very much | 9 | 8
  Hands, 0-Not at all | 100 | 44
  Hands, 1-A little bit | 38 | 24
  Hands, 2-Somewhat | 20 | 19
  Hands, 3-Quite a bit | 17 | 5
  Hands, 4-Very much | 4 | 3
Statistical Analysis 1: Comparison: Non-gBRCA Niraparib vs Non-gBRCA Placebo; Test type: Superiority; p = 0.5037, Pearson's Chi-squared test; Analysis for gBRCA Niraparib vs gBRCA Placebo-Feet
Statistical Analysis 2: Comparison: Non-gBRCA Niraparib vs Non-gBRCA Placebo; Test type: Superiority; p = 0.1640, Pearson's Chi-squared test; Analysis for gBRCA Niraparib vs gBRCA Placebo-Hands

37. Secondary Outcome: Number of Participants With Response to Neuropathy Questionnaire in Cohort With no Germline BRCA at Cycle 4
Description: as for outcome 31
Time Frame: At Cycle 4 (Each cycle was of 28 days)
Population: Intent-to-treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-gBRCA Niraparib | Non-gBRCA Placebo
Number analyzed (Participants) | 181 | 95
Participants
  Feet, 0-Not at all | 54 | 31
  Feet, 1-A little bit | 37 | 16
  Feet, 2-Somewhat | 34 | 17
  Feet, 3-Quite a bit | 20 | 11
  Feet, 4-Very much | 9 | 5
  Hands, 0-Not at all | 89 | 43
  Hands, 1-A little bit | 29 | 21
  Hands, 2-Somewhat | 14 | 10
  Hands, 3-Quite a bit | 14 | 3
  Hands, 4-Very much | 6 | 1
Statistical Analysis 1: Comparison: Non-gBRCA Niraparib vs Non-gBRCA Placebo; Test type: Superiority; p = 0.9599, Pearson's Chi-squared test; Analysis for gBRCA Niraparib vs gBRCA Placebo-Feet
Statistical Analysis 2: Comparison: Non-gBRCA Niraparib vs Non-gBRCA Placebo; Test type: Superiority; p = 0.2470, Pearson's Chi-squared test; Analysis for gBRCA Niraparib vs gBRCA Placebo-Hands

38. Secondary Outcome: Number of Participants With Response to Neuropathy Questionnaire in Cohort With no Germline BRCA at Cycle 6
Description: as for outcome 31
Time Frame: At Cycle 6 (Each cycle was of 28 days)
Population: Intent-to-treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-gBRCA Niraparib | Non-gBRCA Placebo
Number analyzed (Participants) | 144 | 56
Participants
  Feet, 0-Not at all | 43 | 16
  Feet, 1-A little bit | 29 | 10
  Feet, 2-Somewhat | 30 | 11
  Feet, 3-Quite a bit | 18 | 9
  Feet, 4-Very much | 5 | 5
  Hands, 0-Not at all | 68 | 29
  Hands, 1-A little bit | 30 | 10
  Hands, 2-Somewhat | 13 | 6
  Hands, 3-Quite a bit | 9 | 5
  Hands, 4-Very much | 3 | 0
Statistical Analysis 1: Comparison: Non-gBRCA Niraparib vs Non-gBRCA Placebo; Test type: Superiority; p = 0.5921, Pearson's Chi-squared test; Analysis for gBRCA Niraparib vs gBRCA Placebo-Feet
Statistical Analysis 2: Comparison: Non-gBRCA Niraparib vs Non-gBRCA Placebo; Test type: Superiority; p = 0.7459, Pearson's Chi-squared test; Analysis for gBRCA Niraparib vs gBRCA Placebo-Hands

39. Secondary Outcome: Number of Participants With Response to Neuropathy Questionnaire in Cohort With no Germline BRCA at Post-progression
Description: as for outcome 31
Time Frame: Up to 7 years, 7 months and 4 days
Population: Intent-to-treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-gBRCA Niraparib | Non-gBRCA Placebo
Number analyzed (Participants) | 185 | 105
Participants
  Feet, 0-Not at all | 57 | 32
  Feet, 1-A little bit | 45 | 12
  Feet, 2-Somewhat | 23 | 16
  Feet, 3-Quite a bit | 19 | 16
  Feet, 4-Very much | 5 | 8
  Hands, 0-Not at all | 88 | 48
  Hands, 1-A little bit | 35 | 15
  Hands, 2-Somewhat | 13 | 9
  Hands, 3-Quite a bit | 7 | 10
  Hands, 4-Very much | 3 | 1
Statistical Analysis 1: Comparison: Non-gBRCA Niraparib vs Non-gBRCA Placebo; Test type: Superiority; p = 0.0259, Pearson's Chi-squared test
Statistical Analysis 2: Comparison: Non-gBRCA Niraparib vs Non-gBRCA Placebo; Test type: Superiority; p = 0.2798, Pearson's Chi-squared test; Analysis for gBRCA Niraparib vs gBRCA Placebo-Hands

40. Secondary Outcome: Number of Participants With Concordance of a Candidate Companion BRAC Analysis Diagnostic Test Compared to the Centralized BRCA Mutation Test Used in This Study
Description: This will never be analyzed since the data for the candidate companion BRAC analysis diagnostic test was not collected which was to be compared with centralized BRCA mutation test used in this study.
Time Frame: Up to 7 years, 7 months and 4 days
Population: Intent-to-treat Population.
Arm/Group | gBRCA Niraparib | gBRCA Placebo
Number analyzed (Participants) | 0 | 0

41. Secondary Outcome: Number of Participants With Concordance of a Candidate Companion HRD Diagnostic Test Compared to the HRD Test Used in This Study
Description: This will never be analyzed since the data for the candidate companion HRD diagnostic test was not collected which was to be compared with HRD test used in this study.
Time Frame: Up to 7 years, 7 months and 4 days
Population: Intent-to-treat Population.
Arm/Group | Non-gBRCA Niraparib | Non-gBRCA Placebo
Number analyzed (Participants) | 0 | 0

42. Secondary Outcome: Number of Participants With Non-serious Adverse Events (AEs) and Serious AEs (SAEs)
Description: An AE is any untoward medical occurrence that occurs in a participants or clinical investigation participant administered a pharmaceutical product, and which does not necessarily have to have a causal relationship with this treatment. A SAE is defined as any untoward medical occurrence that at any dose which results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, is an important medical event(s) as per medical and scientific judgment. Adverse events which were not serious adverse events were considered as non serious adverse events. Data presented for this outcome measure is based on the data cut-off date of 31-March-2021, which aligns with the time of the study unblinding.
Time Frame: Up to 7 years, 7 months and 6 days
Population: Safety Population consisted of all participants who ingested any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | gBRCA Niraparib | gBRCA Placebo | Non-gBRCA Niraparib | Non-gBRCA Placebo
Number analyzed (Participants) | 136 | 65 | 231 | 114
Participants
  Non-serious AEs | 136 | 62 | 231 | 110
  SAEs | 51 | 9 | 76 | 20

43. Secondary Outcome: Number of Participants With Non-serious AEs and SAEs (Post-study Unblinding)
Description: An AE is any untoward medical occurrence that occurs in a participants or clinical investigation participant administered a pharmaceutical product, and which does not necessarily have to have a causal relationship with this treatment. A SAE is defined as any untoward medical occurrence that at any dose which results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, is an important medical event(s) as per medical and scientific judgment. Adverse events which were not serious adverse events were considered as non serious adverse events. The data is presented for post-study unblinding duration 01-Apr-2021 to 26-Dec-2021
Time Frame: Up to 8 months, 26 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Groups:
- gBRCA Niraparib (PSU): Participants with germline breast cancer gene (gBRCA) mutation received oral dose of niraparib 300 milligrams (mg) once daily in 28-day cycles until disease progression. This arm presents data for post-study unblinding duration 1-Apr-2021 to 26-Dec-2021.
Arm/Group | gBRCA Niraparib (PSU) | gBRCA Placebo (PSU) | Non-gBRCA Niraparib (PSU) | Non-gBRCA Placebo (PSU)
Number analyzed (Participants) | 22 | 8 | 31 | 13
Participants
  Non-serious AEs | 0 | 0 | 0 | 0
  SAEs | 0 | 0 | 0 | 0

44. Secondary Outcome: Number of Participants With Non-serious AEs and SAEs in FE Sub-study
Description: An AE is any untoward medical occurrence that occurs in a participants or clinical investigation participant administered a pharmaceutical product, and which does not necessarily have to have a causal relationship with this treatment. A SAE is defined as any untoward medical occurrence that at any dose which results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, is an important medical event(s) as per medical and scientific judgment. Adverse events which were not serious adverse events were considered as non serious adverse events.
Time Frame: Up to 2 years, 3 months and 11 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- FE Niraparib Fasted: Participants received Niraparib 300 mg in fasted condition
- FE Niraparib Fed: Participants received Niraparib 300 mg in fed condition
Arm/Group | FE Niraparib Fasted | FE Niraparib Fed
Number analyzed (Participants) | 16 | 16
Participants
  Non-serious AEs | 4 | 6
  SAEs | 1 | 0

45. Secondary Outcome: Number of Participants With Non-serious AEs and SAEs in QTc Sub-study
Description: as for outcome 44
Time Frame: Up to 5 years 10 months and 22 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | QTc Sub-study: Niraparib
Number analyzed (Participants) | 26
Participants
  Non-serious AEs | 24
  SAEs | 12

46. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC[0-infinity]) Following Administration of Niraparib (FE Sub-study)
Description: Blood samples were collected at indicated time points to analyze AUC(0-infinity) of niraparib.
Time Frame: Pre-dose and at 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post dose
Population: Pharmacokinetic population consisted of all participants who received at least one dose of study drug, with sufficient data available to calculate parameters. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms*hour per milliliter
Arm/Group | FE Niraparib Fasted | FE Niraparib Fed
Number analyzed (Participants) | 15 | 14
Nanograms*hour per milliliter | 29016.1 (18405.23) | 31194 (16894.88)
Statistical Analysis 1: Comparison: FE Niraparib Fasted vs FE Niraparib Fed; Test type: Superiority; Ratio of Least square mean = 1.10, 90% CI 2-sided [0.997 to 1.216]

47. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to the Last Quantifiable Concentration (AUC[0-last]) Following Administration of Niraparib (FE Sub-study)
Description: Blood samples were collected at indicated time points to analyze the AUC(0-last) of niraparib.
Time Frame: Pre-dose (Day -1) and at 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post dose
Population: Pharmacokinetic population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms*hour per milliliter
Arm/Group | FE Niraparib Fasted | FE Niraparib Fed
Number analyzed (Participants) | 16 | 15
Nanograms*hour per milliliter | 28638.1 (17911.86) | 27186.4 (14111.37)
Statistical Analysis 1: Comparison: FE Niraparib Fasted vs FE Niraparib Fed; Test type: Superiority; Ratio of Least square mean = 1.068, 90% CI 2-sided [0.978 to 1.166]

48. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) Following Administration of Niraparib (FE Sub-study)
Description: Blood samples were collected at indicated time points to analyze the maximum observed plasma concentration of niraparib.
Time Frame: Pre-dose (Day -1) and at 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post dose
Population: Pharmacokinetic population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | FE Niraparib Fasted | FE Niraparib Fed
Number analyzed (Participants) | 16 | 15
Nanograms per milliliter | 803.7 (403.35) | 582.1 (228.57)
Statistical Analysis 1: Comparison: FE Niraparib Fasted vs FE Niraparib Fed; Test type: Superiority; Ratio of Least square mean = 0.785, 90% CI 2-sided [0.695 to 0.886]

49. Secondary Outcome: Time to Reach Maximum (Tmax) Following Administration of Niraparib (FE Sub-study)
Description: Blood samples were collected at indicated time points to analyze the tmax of niraparib.
Time Frame: Pre-dose (Day -1) and at 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post dose
Population: Pharmacokinetic population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hour
Arm/Group | FE Niraparib Fasted | FE Niraparib Fed
Number analyzed (Participants) | 16 | 15
Hour | 3.1 [1.7 to 6.1] | 6.1 [1.2 to 23]

50. Secondary Outcome: Terminal Elimination Half-life (t1/2) Following Administration of Niraparib (FE Sub-study)
Description: Blood samples were collected at indicated time points to analyze the t1/2 of niraparib.
Time Frame: Pre-dose (Day -1) and at 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post dose
Population: Pharmacokinetic population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | FE Niraparib Fasted | FE Niraparib Fed
Number analyzed (Participants) | 16 | 14
Hour | 50.5 (17.87) | 47.9 (17.54)

51. Secondary Outcome: Number of Participants With Maximum Post-Baseline QT Interval Corrected by Fridericia's Formula (QTcF) Greater Than Pre-specified Thresholds
Description: 12-lead electrocardiogram was obtained at indicated time points using an automated electrocardiogram machine that measured QTcF interval. The number of participants with maximum post-Baseline ECG value exceeding the following limits have been reported: QTcF interval >450 and <= 480 milliseconds (msec) and >500 msec.
Time Frame: At Baseline (Cycle 1 Day 1, each cycle was of 28 days)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | QTc Sub-study: Niraparib
Number analyzed (Participants) | 26
Participants
  >450 msec | 2
  >480 msec | 0
  >500 msec | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious AEs (non-SAEs) and SAEs were collected up to 8 years, 6 months and 6 days
Description: Safety Population was used to assess SAEs and non-SAEs, which comprised of all participants who ingested any amount of study drug. The data is presented in separate arms for adverse events before unblinding (data cut-off date of 31-March-2021) and post-study unblinding until the end of study (01-April-2021 to 26-December-2021).
Arm/Group | gBRCA Niraparib | gBRCA Placebo | Non-gBRCA Niraparib | Non-gBRCA Placebo | FE Niraparib Fasted | FE Niraparib Fed | QTc Sub-study: Niraparib | gBRCA Niraparib (Post-study Unblinding [PSU]) | gBRCA Placebo (PSU) | Non-gBRCA Niraparib (PSU) | Non-gBRCA Placebo (PSU)
All-Cause Mortality (participants affected / at risk) | 72/136 | 29/65 | 146/231 | 68/114 | 0/16 | 0/16 | 5/26 | 0/22 | 0/8 | 0/31 | 0/13
Serious Adverse Events (participants affected / at risk) | 51/136 | 9/65 | 76/231 | 20/114 | 1/16 | 0/16 | 12/26 | 0/22 | 0/8 | 0/31 | 0/13
Other Adverse Events (participants affected / at risk) | 136/136 | 62/65 | 231/231 | 110/114 | 4/16 | 6/16 | 24/26 | 0/22 | 0/8 | 0/31 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | gBRCA Niraparib (N=136) | gBRCA Placebo (N=65) | Non-gBRCA Niraparib (N=231) | Non-gBRCA Placebo (N=114) | FE Niraparib Fasted (N=16) | FE Niraparib Fed (N=16) | QTc Sub-study: Niraparib (N=26) | gBRCA Niraparib (Post-study Unblinding [PSU]) (N=22) | gBRCA Placebo (PSU) (N=8) | Non-gBRCA Niraparib (PSU) (N=31) | Non-gBRCA Placebo (PSU) (N=13)
Thrombocytopenia (Blood and lymphatic system disorders) | 18 (38) | 0 (0) | 23 (36) | 0 (0) | 0 (0) | 0 (0) | 3 (9) | 0 (0) | 0 (0) | 0 (0) | 0/12 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (6) | 0 (0) | 13 (15) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 0 (0) | 6 (7) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/12 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute erythroid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Behaviour disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Undifferentiated sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactoid reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis in device (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Product use complaint (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | gBRCA Niraparib (N=136) | gBRCA Placebo (N=65) | Non-gBRCA Niraparib (N=231) | Non-gBRCA Placebo (N=114) | FE Niraparib Fasted (N=16) | FE Niraparib Fed (N=16) | QTc Sub-study: Niraparib (N=26) | gBRCA Niraparib (Post-study Unblinding [PSU]) (N=22) | gBRCA Placebo (PSU) (N=8) | Non-gBRCA Niraparib (PSU) (N=31) | Non-gBRCA Placebo (PSU) (N=13)
Anaemia (Blood and lymphatic system disorders) | 74 (259) | 5 (5) | 111 (328) | 7 (11) | 1 (1) | 0 (0) | 12 (23) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 24 (77) | 3 (7) | 42 (128) | 3 (14) | 0 (0) | 0 (0) | 10 (19) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 13 (226) | 2 (3) | 93 (256) | 4 (4) | 0/0 (0) | 0/0 (0) | 13 (36) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 34 (50) | 17 (24) | 63 (93) | 39 (50) | 0 (0) | 0 (0) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 56 (105) | 12 (14) | 96 (163) | 23 (30) | 0 (0) | 1 (1) | 9 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 40 (71) | 15 (28) | 44 (76) | 23 (34) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 7 (9) | 3 (3) | 12 (17) | 9 (10) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 106 (205) | 23 (46) | 168 (304) | 41 (59) | 0 (0) | 0 (0) | 13 (16) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 5 (5) | 4 (4) | 11 (18) | 7 (11) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 57 (96) | 10 (13) | 74 (126) | 21 (31) | 0 (0) | 1 (1) | 10 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 66 (134) | 19 (37) | 110 (189) | 38 (53) | 0 (0) | 1 (1) | 13 (20) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 12 (15) | 2 (3) | 15 (23) | 6 (10) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 20 (25) | 6 (11) | 26 (40) | 5 (5) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 11 (29) | 3 (4) | 15 (32) | 3 (3) | 1 (1) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 7 (17) | 3 (3) | 20 (48) | 5 (9) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 23 (64) | 3 (5) | 31 (79) | 2 (2) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 34 (85) | 1 (1) | 45 (132) | 2 (2) | 0 (0) | 0 (0) | 3 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 20 (42) | 5 (14) | 22 (64) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 30 (49) | 9 (12) | 67 (94) | 18 (22) | 1 (1) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (8) | 5 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 11 (14) | 5 (10) | 15 (26) | 4 (5) | 1 (1) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 15 (40) | 8 (18) | 18 (28) | 6 (14) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 26 (39) | 7 (14) | 43 (53) | 9 (12) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 52 (76) | 7 (12) | 52 (97) | 14 (21) | 0 (0) | 0 (0) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 13 (17) | 4 (4) | 14 (19) | 8 (9) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 26 (36) | 6 (7) | 67 (88) | 10 (11) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 26 (36) | 2 (4) | 42 (60) | 8 (9) | 1 (1) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 (34) | 3 (4) | 49 (62) | 12 (14) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 14 (16) | 1 (1) | 16 (20) | 5 (5) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 38 (123) | 5 (6) | 46 (207) | 4 (5) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 12 (13) | 1 (1) | 14 (18) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 17 (26) | 9 (12) | 24 (36) | 9 (17) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 4 (6) | 6 (7) | 23 (29) | 15 (17) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 23 (37) | 10 (11) | 22 (25) | 9 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 19 (38) | 2/6 (5) | 19 (27) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 27 (75) | 3 (3) | 36 (81) | 13 (17) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 11 (17) | 4 (5) | 16 (23) | 7 (8) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 8 (11) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 7 (9) | 1 (1) | 19 (23) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 11 (38) | 4 (6) | 17 (52) | 5 (17) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 11 (31) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 21 (33) | 4 (7) | 29 (40) | 11 (17) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 15 (18) | 3 (5) | 14 (18) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 10 (13) | 1 (1) | 15 (19) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 6 (8) | 4 (4) | 15 (19) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 9 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 7 (10) | 0 (0) | 13 (21) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 7 (15) | 0 (0) | 15 (27) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 13 (19) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 (44) | 10 (11) | 27 (40) | 14 (20) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 29 (40) | 9 (9) | 33 (38) | 16 (38) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 (27) | 4 (4) | 16 (19) | 13 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 16 (24) | 2 (2) | 14 (15) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 15 (18) | 6 (7) | 21 (24) | 12 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 (14) | 2 (2) | 12 (23) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 8 (9) | 7 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 15 (17) | 6 (6) | 20 (21) | 8 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (13) | 3 (3) | 5 (5) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 11 (13) | 0 (0) | 25 (37) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 9 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 (19) | 2 (2) | 16 (21) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 0 (0) | 12 (15) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 10 (11) | 3 (3) | 24 (43) | 6 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 12 (27) | 7 (11) | 21 (27) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 9 (14) | 2 (3) | 14 (21) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0
Contusion (Injury, poisoning and procedural complications) | 10 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 7 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 14 (19) | 1 (1) | 27 (35) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 11 (13) | 1 (1) | 14 (20) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 7 (11) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 18 (30) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 7 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 22 (25) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-01-29): https://cdn.clinicaltrials.gov/large-docs/74/NCT01847274/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT01847274/SAP_001.pdf